CLINICAL TRIAL: NCT00929669
Title: Effect of Pasireotide LAR on Gonadotroph Adenomas: A Pilot Study
Brief Title: Effect of Pasireotide Long Acting Release (LAR) on Gonadotroph Adenomas
Acronym: LAR
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: unable to identify a third subject
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 809652
Record Dates: First submitted 2009-06-23; First posted 2009-06-29 (Estimated); Results first posted 2017-11-28 (Actual); Last update posted 2017-11-28 (Actual); Status verified 2017-10

CONDITIONS: Gonadotroph Adenomas
Keywords: pituitary tumor; endocrine
MeSH Terms: conditions — Pituitary Neoplasms | interventions — pasireotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pasireotide LAR (Experimental): 80 mg IM once monthly
  Interventions: Drug: pasireotide LAR

INTERVENTIONS:
Drug: pasireotide LAR — pasireotide LAR 80 mg IM once a month
  Other Names: SOM230

SUMMARY:
The purpose of this study is to determine if administration of pasireotide LAR for one year to three patients with gonadotroph adenomas and elevated serum FSH concentrations will reduce the serum follicle-stimulating hormone (FSH) to normal and reduce the adenoma size.

DETAILED DESCRIPTION:
Gonadotroph adenomas are the most common pituitary macroadenomas. Currently no medical treatment as been found that decreases the size of these adenomas, so surgery is the only treatment. The reason to think that pasireotide might affect gonadotroph adenomas is that pasireotide binds avidly to somatostatin subtype 5 receptors, and gonadotroph adenomas express these receptors. For this study, three subjects who have gonadotroph adenomas, as judged by a macroadenoma of the pituitary and elevated serum FSH concentration, will be treated with a long-acting form of pasireotide once a month for one year. The effect of pasireotide on the size of the adenoma will be determined by MRI, and FSH secretion will be judged by the serum concentration.

ELIGIBILITY:
Inclusion Criteria:

* gonadotroph adenoma

Exclusion Criteria:

* visual impairment attributable to the adenoma
* radiation therapy
* active gallbladder disease
* uncontrolled diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2009-06; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter J. Snyder, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was initiated in 6/09 and was terminated in 6/10. 2 subjects were enrolled and 1 subject completed the 12 mos. of the study.
Period: Overall Study
Arm/Group | Pasireotide LAR
Started | 2
Completed | 1
Not Completed | 1
Not completed — elevated glucose levels | 1

BASELINE CHARACTERISTICS:
Arm/Group | Pasireotide LAR
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 2
patients with a gonadotroph adenoma [Number; unit: participants] | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Change in Size of the Adenoma by ≥3 mm in at Least Two Dimensions as Determined by MRI
Description: MRI of the pituitary will be performed at baseline, Month 6 and Month 12 to demonstrate a decrease of ≥3 mm in at least two of three dimensions on MRI (cephalocaudal, transverse, and posterior-anterior). The outcome measure is defined as the number of participants who demonstrated a ≥3 mm decrease in adenoma size in two dimensions.
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | Pasireotide LAR
Number analyzed (Participants) | 1
participants | 0

2. Secondary Outcome: Number of Participants With Change in Serum FSH Concentration (mIU/mL) in Patients Who Have Gonadotroph Adenomas Treated With Pasireotide.
Description: Serum FSH (mIU/mL) will be measured at baseline and then monthly for the 12 months of the study to determine if serum FSH concentrations decrease by 20%.
Time Frame: 12 months
Measure: Number; unit: number of participants
Arm/Group | Pasireotide LAR
Number analyzed (Participants) | 1
number of participants | 0

ADVERSE EVENTS:
Arm/Group | Pasireotide LAR
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pasireotide LAR (N=2)
hyperglycemia (Endocrine disorders) | 2 (2)
elevated liver enzymes (Hepatobiliary disorders) | 1 (1)
sinus bradycardia (Cardiac disorders) | 1
pain radiating down leg (Musculoskeletal and connective tissue disorders) | 1
photophobia (Eye disorders) | 1

LIMITATIONS AND CAVEATS:
This trial was terminated due to difficulty in identifying 3 subjects for completion of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes